CLINICAL TRIAL: NCT03046992
Title: A Phase I/II, Open-Label, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Anti-Tumor Activity of YH25448 in Patients with EGFR Mutation Positive Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Clinical Trial of YH25448 in Patients with EGFR Mutation Positive Advanced NSCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YH25448-201
Record Dates: First submitted 2017-01-26; First posted 2017-02-08 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2023-04

CONDITIONS: EGFR Gene Mutation
Keywords: EGFR; Non-Small Cell Lung Cancer; T790M; Brain Metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- YH25448 (Experimental): * Dose Escalation Phase: Consists of 7 Cohorts
  * Dose Expansion Phase: Consists of 5 Cohorts
  * Dose Extension Phase: Consists of 2 Cohorts
  Interventions: Drug: YH25448

INTERVENTIONS:
Drug: YH25448 — * Dose Escalation: YH25448 20mg~320mg, PO
  * Dose Expansion: YH25448 40mg~240mg, PO
  * Dose Extension: Recommended Dose 240mg of YH25448

SUMMARY:
YH25448 is an oral, highly potent, mutant-selective and irreversible EGFR Tyrosine-kinase inhibitors (TKIs) targets both the T790M mutation and activating EGFR mutations while sparing wild type-EGFR. YH25448 is expected to beneficial for the NSCLC patients with brain metastasis due to good blood brain barrier (BBB) penetration property as well as for the treatment of primary lung lesion and extracranial lesions. This study will be conducted to evaluate the safety, tolerability and efficacy of YH25448 in locally advanced or metastatic NSCLC patients with EGFR mutations.

DETAILED DESCRIPTION:
This is a first time in patient study primarily designed to evaluate the safety, tolerability, and efficacy of YH25448 in in patients with EGFR mutation positive (EGFRm+) advanced NSCLC with or without asymptomatic brain metastasis who progressed following prior therapy with an EGFR TKIs agent. This study is composed of 3 parts; part A is a dose escalation phase, part B is a dose expansion phase and part C is a dose extension phase.

In dose escalation phase, YH25448 will be escalated to reach either a maximum tolerated or absorbable dose in patients as defined by dose-limiting toxicity in NSCLC patients who progressed following prior EGFR TKIs treatment to evaluate the safety and tolerability. In dose expansion phase, further safety, tolerability, pharmacokinetic(PK) and efficacy will be evaluated at each dose level(s) of dose escalation phase in NSCLC patients who progressed following prior EGFR TKIs treatment and harbouring confirmed T790M mutation. In dose extension phase, additional 2 cohorts (2nd line therapy cohort, 1st line therapy cohort) will be enrolled to further assess the efficacy, safety, tolerability, and PK of YH25448 at the maximum tolerated dose (MTD) or recommended dose (RD) defined through dose escalation phase and dose expansion phase. Results of these studies will serve as the evidence for further clinical development.

This study will also characterize the metabolite(s) profile of YH25448 and determine PK of its metabolite(s) in biological samples if necessary. Also, exploratory correlation between biomarker profiles and pharmacokinetics/pharmacodynamics will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of NSCLC with single activating EGFR mutations.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 3 months.
* At least one measurable extracranial lesion, not previously irradiated and not chosen biopsy during the study screening period.
* Prior to enrolling in the study, patients must have central confirmation of T790M+ mutation status from a sample taken after documented progression on the EGFR-TKIs therapy according to cohort.

Exclusion Criteria:

* Spinal cord compression.
* Brain metastases with symptomatic and/or requiring steroid for at least 2 weeks prior to start of study treatment.
* Known intracranial hemorrhage which is unrelated to tumor.
* Central Nervous System (CNS) complications that require urgent neurosurgical intervention (e.g. resection or shunt placement).
* Leptomeningeal metastasis prior to study treatment.
* Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
* Any cardiovascular disease as followed.

  * History of symptomatic congestive heart failure (CHF) or serious cardiac arrhythmia requiring treatment
  * History of myocardial infarction or unstable angina within 6 months of the first dose of study treatment
  * Left ventricular ejection fraction (LVEF) < 50%

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability by Common Terminology Criteria for Adverse Events (CTCAE) v4.03 | Safety and tolerability profile will be collected from baseline until 28 days after the last dose, expected average 1 year.
  To assess the safety and tolerability profile of YH25448 by Common Terminology Criteria for Adverse Events (CTCAE) v4.03; vital signs (blood pressure, pulse, weight); laboratory parameters (clinical chemistry, hematology, urinalysis); physical examination; centrally reviewed electrocardiograms (ECGs), echocardiogram or multiple gated acquisition scan and performance status.
Objective Response Rate (ORR) | At baseline and every 6 weeks from first dose objective disease progression or withdrawal from study, up to approximately 1 year.
  Per Response Evaluation Criteria in Solid Tumours (RECIST version 1.1) assessed by MRI or CT. ORR is the percentage of patients with at least 1 visit response of Complete Response (CR) or Partial Response (PR) (according to independent review), prior to progression or further anti-cancer therapy.

SECONDARY OUTCOMES:
Duration of Response (DoR) | At baseline and every 6 weeks from first dose objective disease progression or withdrawal from study, up to approximately 1 year.
  Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT.
Disease Control Rate (DCR) | At baseline and every 6 weeks from first dose objective disease progression or withdrawal from study, up to approximately 1 year.
  Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT.
Progression-Free Survival (PFS) | At baseline and every 6 weeks from first dose objective disease progression or withdrawal from study, up to approximately 1 year.
  Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT. Kaplan-Meier plots will be used to summarize the progression-free survival.
Overall Survival (OS) | At baseline and every 6 weeks from first dose objective disease progression or withdrawal from study, up to approximately 1 year.
  To obtain assessment of anti-tumor activity of YH25448 by evaluation of tumor response using RECIST version 1.1.
Tumor shrinkage | At baseline and every 6 weeks from first dose objective disease progression or withdrawal from study, up to approximately 1 year.
  To obtain assessment of anti-tumor activity of YH25448 by evaluation of tumor response using RECIST version 1.1.
Objective Intracranial Response Rate (OIRR) | At baseline and every 6 weeks from first dose objective disease progression or withdrawal from study, up to approximately 1 year.
  To obtain assessment of anti-tumor activity of YH25448 by evaluation of tumor response using RECIST version 1.1.
Duration of Intracranial Response (DoIR) | At baseline and every 6 weeks from first dose objective disease progression or withdrawal from study, up to approximately 1 year.
  To obtain assessment of anti-tumor activity of YH25448 by evaluation of tumor response using RECIST version 1.1.
Intracranial Progression Free Survival (IPFS). | At baseline and every 6 weeks from first dose objective disease progression or withdrawal from study, up to approximately 1 year.
  To obtain assessment of anti-tumor activity of YH25448 by evaluation of tumor response using RECIST version 1.1. Kaplan-Meier plots will be used to summarize the progression-free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Yuhan Corporation, Study Director — Clinical Development Department
Locations (16):
- South Korea (16):
  - The Catholic University of Korea, Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Inje University Haeundae Paik Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Severance Hospital, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han JY, Ahn MJ, Lee KH, Lee YG, Kim DW, Min YJ, Kim SW, Cho EK, Kim JH, Lee GW, Lee SS, Lee NM, Jang HW, Han H, Park H, Lee J, Cho BC. Updated overall survival and ctDNA analysis in patients with EGFR T790M-positive advanced non-small cell lung cancer treated with lazertinib in the phase 1/2 LASER201 study. BMC Med. 2024 Oct 8;22(1):428. doi: 10.1186/s12916-024-03620-8. PMID 39379931
- [Derived] Kim B, Lee J, Jang H, Lee N, Mehta J, Jang SB. Effects of Acid-Reducing Agents on the Pharmacokinetics of Lazertinib in Patients with EGFR Mutation-Positive Advanced Non-Small-Cell Lung Cancer. Adv Ther. 2022 Oct;39(10):4757-4771. doi: 10.1007/s12325-022-02286-z. Epub 2022 Aug 13. PMID 35962934
- [Derived] Cho BC, Han JY, Kim SW, Lee KH, Cho EK, Lee YG, Kim DW, Kim JH, Lee GW, Lee JS, Shim BY, Kim JS, Chun SH, Lee SS, Kim HR, Hong MH, Ahn JS, Sun JM, Lee Y, Lee DH, Kang JA, Lee N, Kwon MJ, Espenschied C, Yablonovitch A, Ahn MJ. A Phase 1/2 Study of Lazertinib 240 mg in Patients With Advanced EGFR T790M-Positive NSCLC After Previous EGFR Tyrosine Kinase Inhibitors. J Thorac Oncol. 2022 Apr;17(4):558-567. doi: 10.1016/j.jtho.2021.11.025. Epub 2021 Dec 24. PMID 34958928
- [Derived] Ahn MJ, Han JY, Lee KH, Kim SW, Kim DW, Lee YG, Cho EK, Kim JH, Lee GW, Lee JS, Min YJ, Kim JS, Lee SS, Kim HR, Hong MH, Ahn JS, Sun JM, Kim HT, Lee DH, Kim S, Cho BC. Lazertinib in patients with EGFR mutation-positive advanced non-small-cell lung cancer: results from the dose escalation and dose expansion parts of a first-in-human, open-label, multicentre, phase 1-2 study. Lancet Oncol. 2019 Dec;20(12):1681-1690. doi: 10.1016/S1470-2045(19)30504-2. Epub 2019 Oct 3. PMID 31587882
- [Derived] Yun J, Hong MH, Kim SY, Park CW, Kim S, Yun MR, Kang HN, Pyo KH, Lee SS, Koh JS, Song HJ, Kim DK, Lee YS, Oh SW, Choi S, Kim HR, Cho BC. YH25448, an Irreversible EGFR-TKI with Potent Intracranial Activity in EGFR Mutant Non-Small Cell Lung Cancer. Clin Cancer Res. 2019 Apr 15;25(8):2575-2587. doi: 10.1158/1078-0432.CCR-18-2906. Epub 2019 Jan 22. PMID 30670498